CLINICAL TRIAL: NCT05789472
Title: The Relationship Between Reaction Time and Executive Functions in Amateur Female Athletes Playing Team Sports
Brief Title: The Relationship Between Reaction Time and Executive Functions in Female Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Gülay Aras, Principal Investigator, Medipol University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 119
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Assessment
Keywords: Female Athlete; Executive Function; Reaction Time
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Football Group (Experimental): Assessment
  Interventions: Behavioral: Assessment
- Basketball Group (Experimental): Assessment
  Interventions: Behavioral: Assessment
- Volleyball Group (Experimental): Assessment
  Interventions: Behavioral: Assessment

INTERVENTIONS:
Behavioral: Assessment — Executive functions and reaction times of all participants will be measured.

SUMMARY:
The literature shows the positive effects of regular physical activity and sports on executive functions. It is seen that the low reaction times of the athletes increase their success and prevent injuries. However, as a result of the examinations, no studies were found that examined the relationship between the reaction times of the athletes and their executive functions. In this context, it is aimed to examine the relationship between reaction time and executive functions in amateur female athletes who play team sports.

DETAILED DESCRIPTION:
Executive functions are often described as 'higher cognitive processes' that govern other basic cognitive functions. Executive functions include higher-order cognitive abilities such as planning, decision making, problem solving, strategizing, working memory, inhibition, cognitive flexibility, abstraction, and reasoning. It enables individuals to organize their thoughts and actions during goal-directed behavior, to think, to produce ideas, to respond and to control in the face of unexpected situations.

Response time is the time elapsed after the stimulus reaches the body until the first response to these stimuli. It is the time between the first reaction that occurs after the appearance of a sensory, visual or tactile stimulus. Athletes must respond quickly to a ball, the movement of another athlete, or incoming signals to compete successfully and avoid injury. The reaction time depends on the neurophysiological processes in the brain.

In our study, which was planned to evaluate the relationship between reaction time and executive functions in 66 amateur female athletes between the ages of 18-25, who are university football, basketball and volleyball team athletes; The age, body mass index (BMI), sports branch, duration of interest in sports will be recorded in the demographic information form. Hand-eye and foot-eye reaction time of the athletes will be evaluated by BlazePod Reaction Time Determination Test and executive functions will be evaluated with Forward-Backward Number Range test, Stroop test and Tracking A-B test.

ELIGIBILITY:
Inclusion Criteria:

* At least 5 years of sports
* Being an athlete on university sports teams

Exclusion Criteria:

* Athletes with health problems (eg cancer, arthritis, heart disease, lung disease, neurological or psychological illness)

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only female
Enrollment: 66 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
BlazePod Reaction Time Determination Test | 1 day
  The BlazePod test, which includes "pods" equipped with touch sensors and LED lights, will be used to evaluate the reaction time.
  In the evaluation, the number of 15 seconds of touch (number), the reaction time (ms) for the visual response of 15 seconds of touch, and the average reaction time will be analyzed.
Forward-Backward Number Range Test | 1 day
  The test consists of two parts as forward and backward range. In the forward number range, the numbers are read at one-second intervals and the patient is asked to repeat the numbers read randomly in the same order. In the back number range, it is requested to repeat the numbers read from the end to the beginning. As you succeed, it continues by increasing one step. If the patient fails twice in a row for both sections, the test is discontinued. Generally, the difference between the forward and backward number range is expected to be two digits. The highest score that can be obtained for the forward range is 8 points, and 7 for the backward range, for a total of 15 points.
Stroop Test | 1 day
  The test consisting of 6 lines of random blue, green, red colors and including three basic tasks; In the first task, the individual is asked to name the colors in the box. In case of successful completion, the second task, the words written with the same colors, is asked to be read and the time is kept. In the third task, the words are asked to inhibit reading and to say in which color they are written. The time to finish the test, the number of errors, and the number of spontaneous corrections are noted.
Tracking Test | 1 day
  The trail riding test consists of two parts, A and B. In part A, the participants are asked to combine the circles with the numbers in the correct order and following each other (1-2-3-4-5...). In section B, there are letters and numbers placed in circles. Participants are asked to combine letters and numbers in the correct sequence (1-A-2-B-3-C-4-D...). The times of both sections are recorded. The trailing test requires visuospatial processing and motor skills. Particularly, part B is widely used in the measurement of complex attention, planning, set-changing, and reaction inhibition among executive functions.

CONTACTS AND LOCATIONS:
Overall Officials: Gülay Aras Bayram, PhD, Principal Investigator — Medipol University
Locations (1):
- Gülay Aras Bayram, Istanbul, Atatürk Street, Turkey (Türkiye)